CLINICAL TRIAL: NCT05459337
Title: Multidisciplinary Support to Access Living Donor Kidney Transplant (MuST AKT)
Acronym: MuST AKT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00121297
Record Dates: First submitted 2022-06-22; First posted 2022-07-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Living Donor Kidney Transplantation

STUDY DESIGN:
Intervention Model Description: Parallel block randomized control trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This arm will receive the MuST AKT intervention, which is a multidisciplinary, tailored person-centered behavioural intervention designed to "help and enable" the potential kidney transplant recipients to achieve what is required to receive a living donor kidney transplantation.
  Interventions: Behavioral: MuST AKT
- Usual Care (control) (No Intervention): In the usual care (control) condition, participants will go through the current standard of care, which is a social worker assessment.

INTERVENTIONS:
Behavioral: MuST AKT — A behavioural intervention designed to help participants identify and communicate with their social network about living kidney donation.
  Arms: Intervention

SUMMARY:
For people living with kidney failure, the two active treatment options are dialysis or kidney transplantation. Transplantation is optimal, and especially from a living donor - offering patients longer survival, a better quality of life, and cost savings for the health system when compared to dialysis. However, 20% of patients die on dialysis while waiting for a deceased donor organ. As the rate of kidney failure continues to rise, the gap between demand and supply of the organs for transplantation increases.

Compared to other provinces in Canada, the rate of living kidney donor transplantation is lower in Alberta, so it is essential that improvements are made to the process around living kidney donor transplantation, for better patient outcomes and care.

Our published evidence-based review on strategies to increase living kidney donation, found that for patients with kidney failure, the intervention with the greatest health impact was personalized support, provided by a multidisciplinary team, to inform and educate the patients' social network. A province-wide survey also confirmed that many patients with kidney failure are unable to find a living kidney donor and also find it difficult to approach potential donors due to lack of skills, supports, and resources.

The investigators have developed the Multidisciplinary Support To Access living donor Kidney Transplant (MuST AKT) intervention to support potential kidney transplant recipients find living donors through their social networks, and thereby increase the number of living kidney donor transplants in Alberta. The investigators will test the effectiveness of this intervention.

DETAILED DESCRIPTION:
Living donor kidney transplantation (LDKT) is the optimal treatment for end-stage kidney disease patients, offering patients longer survival, a better quality of life, and cost savings for the health system when compared to dialysis. Outcome data shows that only 16% of Canadians on dialysis survive past 10 years, whereas up to 74% of Canadians with a kidney transplant have a functioning kidney after 10 years. The ideal treatment trajectory is to avoid dialysis entirely and receive a living donor transplant prior to dialysis (pre-emptive), which unfortunately only occurs in 10.5% of eligible patients.

Patients with kidney failure report barriers to LDKT, including navigating the system, addressing their concerns and fears, identifying and approaching potential living donors, keeping motivated, and then utilizing the ones unable to donate as advocates. To address these barriers and increase LDKT, the MuST AKT intervention has been developed. MuST AKT is designed to provide personalized support and enable potential kidney transplant recipients to communicate their story and desire for a LDKT with their personal and broader social networks.

A definitive Randomized Controlled Trial is proposed to test the effectiveness of the MuST AKT intervention to increase LDKT outcomes in a larger sample, before scaling to and implementing across Alberta.

Primary Objective:

The primary objective of this study is to examine the effectiveness of the MuST AKT intervention to increase living donor kidney transplantation outcomes.

Hypothesis:

The MuST AKT intervention will increase living donor kidney transplant outcomes compared to the control condition (standard care).

Additional Objectives:

The secondary objective is to evaluate patient outcome improvement by collecting Patient Reported Outcome Measures (PROMs) to assess the proportion of patients who find at least one potential living donor.

The tertiary objective is to evaluate patient experience by collecting i) qualitative interviews and ii) Patient Reported Experience Measures (PREMs) to determine whether this program would be recommended to other patients and to what extent this program helped find a potential living kidney donor.

The quaternary objective is to evaluate the feasibility of this program by assessing consent rate, attendance, adherence, drop-out, intervention fidelity, and cost-effectiveness.

Research Methods/Procedures:

This is a definitive parallel randomized controlled trial with a qualitative interview component. The intervention condition will receive a multidisciplinary, tailored person-centered intervention over three months (MuST AKT program), and the control condition will receive the current standard of care (social worker assessment).

Patients who have been referred for kidney transplantation assessment in Edmonton will be contacted during a standard care kidney transplant education session or over the telephone if the education has been completed. Consenting participants meeting the eligibility requirements will be contacted via telephone by a member of the research team to confirm their enrollment and complete a baseline questionnaire to assess socio-demographics and PREMs. Then participants will be randomized to either the intervention or control condition, using predetermined randomly-generated (by Stata MP 15·1) permuted blocks of 4 and 6. Assignment to condition will be concealed by the database up until the point of assignment. All group and individual sessions will be held either virtually or in-person, at the participants discretion, as long as there are no public health (e.g., COVID-19) restrictions that would prevent in-person visits. If there are public health restrictions that prevent in-person visits, the sessions will be held virtually. Consent rate, attendance, adherence, drop-out, and intervention fidelity will be tracked during enrollment and throughout the duration of the intervention. Upon completion of the intervention (or usual care), participants will complete a post-intervention questionnaire to assess PREMs. Participants in the MuST AKT intervention condition who complete the intervention sessions will be contacted to participate in a semi-structured qualitative interview over the telephone (approximately 45 minutes) within two weeks of their last session. Participants who complete the MuST AKT intervention condition but have not had a potential donor come forward after 12 months of the last session will be contacted to complete a semi-structured interview over the telephone (approximately 20 minutes) to explore factors contributing to their lack of success. Kidney transplant status will be tracked for a period of 24 months post-intervention.

The cost-effectiveness of the intervention will be evaluated after participant data collection is complete (24 months), and values obtained from study records (cost of developing and delivering intervention) and previously published estimates of living donor work-ups and transplantation costs, and cost-savings due to forgoing of alternative therapies (i.e., dialysis).

Intervention Condition: MuST AKT is a multidisciplinary, tailored person-centered intervention aimed to support participants identification of potential donors and communication with their social network. An introductory session will be followed by three sessions (all one-on-one) and a final session 4 with participants family and friends (potential donors and advocates) identified in session 1. The introductory session will be approximately 60 minutes and the remaining intervention sessions will be approximately 90 minutes. Sessions will be facilitated by a trained licensed social worker, a coordinator, or a media expert, with extra training in kidney disease, transplantation, living kidney donation, counselling and interviewing, and patient confidentiality.

Usual care (control condition): In the control condition, participants will go through the current standard of care, which is a social worker assessment. If the intervention is successful in the definitive RCT and approved by Alberta Health Services as the 'new standard of care', people in control condition will be contacted and given the option to participate in the MuST AKT intervention.

Additional Interviews with separate informed consent procedures: Friends and family members of participants taking part in session 4 will be invited to participate in a sub-study, which aims to explore their experiences of group session 4. Those expressing interest will be contacted by a qualitative researcher via telephone, and following informed consent, will participate in a semi-structured interview lasting approximately 20 minutes.

Plan for Data Analysis:

Quantitative: All analyses will be completed in Stata/MP 17.0 (www.stata.com), using an intention-to-treat approach. Fisher's exact tests (for dichotomous outcomes), and t-tests or Wilcoxon rank-sum tests (for continuous outcomes data), will be used as appropriate. Unadjusted proportions, means or medians and their differences along with 95% confidence intervals will be reported. P <0.05 will be considered statistically significant for all quantitative outcomes. Residual, leverage and influence diagnostics will be examined.

Our primary analyses (which includes primary and secondary outcomes) will pool data from both the pilot and the current trials. In secondary analyses, we will generate within trial results to investigate potential heterogeneity of intervention delivery.

Qualitative: Data will be analyzed in NVivo-12 by experienced qualitative researchers independent of the study, using deductive thematic analysis. A coding framework will be established based on the interview guides and updated to include additional themes that emerge from the data. The coding framework will be validated by two coders, any disagreements will be resolved through discussion.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* No obvious contraindication to kidney transplantation
* Successfully completed 'introduction to kidney transplant' module

Exclusion Criteria:

* Potential Living Kidney Donor identified
* Previously received organ transplant
* Candidate for multi-organ transplant
* Stanford Integrated Psychosocial Assessment for Transplant (SIPAT) Score >20
* Rapid Estimate of Adult Literacy in Medicine (REALM-66) score <19(illiterate in English)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Living Kidney Donor Transplantation | 24 months
  Proportion of participants undergoing living kidney donor transplantations

SECONDARY OUTCOMES:
Living Kidney Donor Evaluation Approved | 12 months
  Proportion of participants with ≥1 approved LDKT
Living Kidney Donor Evaluation Started | 12 months
  Proportion of participants with at least one donor who started evaluation for living kidney donation
Contact Living Donor Services | 12 months
  Proportion of participants with at least one donor who contacted living donor services

OTHER OUTCOMES:
Consent rate | From start date to end date of study recruitment, up to 1 year
  Proportion of potentially eligible participants who gave consent (consent rate) and reasons for decline of consent.
Reasons for decline of consent | From start date to end date of study recruitment, up to 1 year
  Reasons for decline of consent.
Non-completion of initial screening | From start date to end date of study recruitment, up to 1 year
  Proportion of potential participants who did not complete the initial screening.
Initial screening exclusion | From start date to end date of study recruitment, up to 1 year
  Proportion of potential participants who were excluded after initial screening
Intervention session completion | From date of first to last documented session, an average of 3 months
  Proportion of participants who completed each session of the program.
Drop-out rate (overall study) | From start date to end date of study recruitment, up to 1 year
  Proportion of participants who withdrew consent.
Intervention sessions drop-out (all four) | From date of first to last documented session, an average of 3 months
  Proportion of participants who did not complete all four sessions.
Intervention sessions drop-out (individual sessions) | From date of first to last documented session, an average of 3 months
  Proportions of sessions postponed and not completed.
Session duration | From date of first to last documented session, an average of 3 months
  Actual duration of the intervention period for each participant.
Participant recommendation | At date of last documented session, an average of 3 months
  The proportion of the patients who 'recommend' this program to other patients.
Perception of program effectiveness as assessed by 1 item developed for this study | At date of last documented session, an average of 3 months
  Participants rate the following prompt on a scale from 1(completely disagree) to 7 (completely agree): "This program was effective at finding me a living kidney donor". A higher score indicates a better outcome.
Self-efficacy for approaching a potential donor as assessed by 1 item developed for this study: "How confident are you that you can talk to a friend or family member about being a potential living kidney donor?" | 3 months (length of intervention)
  Participants rate the following prompt on a scale from 0 (not at all confident) to 100 (complete confidence): "How confident are you that you can talk to a friend or family member about being a potential living kidney donor?". Higher scores indicate a better outcome.
Self-efficacy for finding a living kidney donor assessed by 1 item developed for this study: "How confident are you that you can find a potential living kidney donor?" | 3 months (length of intervention)
  Participants rate the following prompt on a scale from 0 (not at all confident) to 100 (complete confidence): "How confident are you that you can find a potential living kidney donor?". Higher scores indicate a better outcome.
Identified donor and advocate | From date of first to last documented session, an average of 3 months
  Proportion of participants who identified at least one potential donor and/or advocate.
Wrote their story | At date of first documented session, an average of 3 months
  Proportion of participants who 'wrote their stories' at the end of session 1.
Conversation started | From date of first to last documented session, an average of 3 months
  Proportion of participants who started a conversation with at least one potential donor.
Friend and family member attendance at the last intervention session | At date of last documented session, an average of 3 months
  Total number of people who attend the last intervention session
Cost-effectiveness | 24 months
  Total cost (including development and delivery of the intervention, donor work-ups, transplantations) minus the cost-savings due to forgoing or stopping dialysis.
Intervention fidelity | From date of first to last documented session, an average of 3 months
  Proportion of session tasks and activities completed by the intervention facilitator.
Contact Living Donor Services (numbers) | 12 months
  The number of potential living donors who contacted living donor services per participant

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shojai, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No